CLINICAL TRIAL: NCT06068101
Title: Clinical and Genetic Investigation of the Association Between Primary Aldosteronism and Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, ANA ALICE WOLF MACIEL, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Other Study IDs: Primary Aldosteronism + Cancer
Record Dates: First submitted 2023-08-15; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Thyroid Cancer, Papillary; Primary Aldosteronism
MeSH Terms: conditions — Thyroid Cancer, Papillary; Hyperaldosteronism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with papillary thyroid cancer (PTC) and EH (essential hypertension): Primary Aldosteronism was investigated in all patients with PTC and EH (n= 137), regardless of hypertension severity, under active surveillance at a cancer institute from 2019 to 2022.
  Interventions: Diagnostic Test: Secreening test for primary aldosteronism and Confirmatory Testing
- Patients with EH (essential hypertension) previously investigated for PA (primary aldosteronism): The control group included 137 (1:1) age,sex and body mass index (BMI) matched individuals from a retrospective cohort of EH previously investigated for PA from 2011 to 2022.

INTERVENTIONS:
Diagnostic Test: Secreening test for primary aldosteronism and Confirmatory Testing — Serum aldosterone and plasma direct renin concentrations were measured by a chemiluminescent immunoassay. A positive PA screening was defined by aldosterone > or = 10 ng/dL and aldosterone to renin ratio > or = 2 ng/dL/uUI/mL
  Groups: Patients with papillary thyroid cancer (PTC) and EH (essential hypertension)

SUMMARY:
Aldosterone excess can cause oxidative stress leading to DNA damage in vitro and in vivo. Single case reports demonstrated a coincidence of primary aldosteronism (PA) with different malignancies. A higher prevalence of thyroid nodules and non-toxic multinodular goiter was described in patients with PA compared to those with essential hypertension (EH). A single study showed an association between PA and papillary thyroid cancer (PTC), but without a paired control group. Objective: To assess PA prevalence in a transversal cohort of patients with PTC and EH compared to a paired control group with HT.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is the most frequent cause of endocrine hypertension, with an estimated prevalence of 20% among individuals with resistant hypertension. PA is associated with an increased risk of malignancy, probably due to aldosterone effects in promoting cell proliferation. Recently, a high prevalence of PA was demonstrated in patients with essential hypertension (EH) and papillary thyroid cancer (PTC), similarly to the prevalence of PA among individuals with resistant EH. In addition, abnormalities in thyroid ultrasound (non-toxic multinodular goiter) are more common in PA patients when compared to controls. Despite of this initial evidence, the link between PA and PTC remains to be elucidated. Then, the aim of this study is to investigate the clinical and genetic aspects of the association between PA and PTC. The specific aims are: 1) To evaluate the prevalence of PA in a transversal cohort of patients with EH and PCT; 2) To investigate thyroid ultrasonography abnormalities in PA patients; 3) To perform exome sequencing (blood DNA) in patients with PA and PTC paired with tumor tissue; and 4) To conduct functional studies of the novel genetic variants identified by exome sequencing. To achieve this goal, the investigators will employ the following techniques: next-generation sequencing, bioinformatic analysis, real-time PCR and immunohistochemistry. In this project, the investigators expect to establish the prevalence of PA among patients with EH and PTC, and to identify new genetic targets involved in the association between PA in PTC.

ELIGIBILITY:
Inclusion Criteria:

* All patients with PTC and EH regardless of hypertension severity

Exclusion Criteria:

* Patients who were using medications that secondarily increase blood pressure levels were excluded
* Did not agree to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this cross-sectional case-control study, PA was investigated in all patients with PTC and EH (n= 137), regardless of hypertension severity, under active surveillance at a cancer institute from 2019 to 2022. The control group included 137 (1:1) age-, sex- and body mass index (BMI)-matched individuals from a retrospective cohort of EH previously investigated for PA from 2011 to 2022. Serum aldosterone and plasma direct renin concentrations were measured by a chemiluminescent immunoassay. A positive PA screening was defined by aldosterone > or = 10 ng/dL and aldosterone to renin ratio > or = 2 ng/dL/uUI/mL.
Sampling Method: Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
PA prevalence in a transversal cohort of patients with PTC and EH | Through study completion, an average of 1,5 year
  To assess PA prevalence in a transversal cohort of patients with PTC and EH compared to a paired control group with EH

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Alice Wolf Maciel, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No